CLINICAL TRIAL: NCT00005971
Title: A Phase II Study of Flavopiridol (HMR 1275; NSC 649890) in Patients With Previously Untreated Metastatic Malignant Melanoma
Brief Title: Flavopiridol in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I137; CAN-NCIC-IND137 (Other: PDQ); NCI-NCIC-137 (Other: NCI); CDR0000067955 (Other: PDQ)
Record Dates: First submitted 2000-07-05; First posted 2003-05-21 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: alvocidib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of flavopiridol in treating patients who have metastatic malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy of flavopiridol in patients with previously untreated metastatic malignant melanoma.
* Assess the toxicity of this treatment in these patients.
* Assess the time to progression, early progression rate, and response duration in these patients when treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive flavopiridol IV over 1 hour on days 1-3. Treatment continues every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, and then every 3 months until disease progression or death.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic malignant melanoma not amenable to standard curative therapies

  * No prior regional or systemic therapy for metastatic disease
* Measurable disease

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Bone lesions not considered measurable
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 2.5 times ULN

Renal:

* Creatinine no greater than ULN

Cardiovascular:

* If history of cardiac disease, ejection fraction greater than 50%
* No clinically significant cardiac symptomology

Pulmonary:

* If history of pulmonary disease, FEV1, FVC, and TLC greater than 60% predicted and DLCO greater than 50% predicted
* No clinically significant pulmonary symptomology

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent serious disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior adjuvant immunotherapy allowed
* No prior immunotherapy for metastatic disease

Chemotherapy:

* No prior chemotherapy for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior adjuvant hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* Must have measurable disease outside irradiated area OR
* Evidence of progression or new lesions in irradiated area
* No more than 25% of functioning bone marrow irradiated
* No concurrent radiotherapy to sole site of measurable disease

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No other concurrent anticancer therapy or investigational anticancer agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2000-07-04 (Actual); Primary Completion 2001-08-24 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Burdette-Radoux, MD, Study Chair — McGill Cancer Centre at McGill University
Locations (50):
- Canada (50):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Lethbridge Cancer Clinic, Lethbridge, Alberta
  - Penticton Regional Hospital, Penticton, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Hamilton and Disrict Urology Association, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - York County Hospital, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Male Health Centre/CMX Research Inc., Oakville, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Scarborough Hospital - General Site, Scarborough Village, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier de l'Universite' de Montreal, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burdette-Radoux S, Tozer RG, Lohmann RC, Quirt I, Ernst DS, Walsh W, Wainman N, Colevas AD, Eisenhauer EA. Phase II trial of flavopiridol, a cyclin dependent kinase inhibitor, in untreated metastatic malignant melanoma. Invest New Drugs. 2004 Aug;22(3):315-22. doi: 10.1023/B:DRUG.0000026258.02846.1c. PMID 15122079
- [Result] Burdette-Radoux S, Tozer RG, Lohmann R, et al.: NCIC CTG phase II study of flavopiridol in patients with previously untreated metastatic malignant melanoma (IND.137). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1382, 2002.